CLINICAL TRIAL: NCT01278680
Title: Incentives for Moving
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment has not begun; study suspended indefinitely due to change in management at company where we were going to conduct the study.
Sponsor: Harvard University (Other)
Collaborators: University of California, Berkeley (Other); Carnegie Mellon University (Other)
Responsible Party: Principal Investigator, Michael Norton, Associate Professor, Harvard University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Walkstation3
Record Dates: First submitted 2011-01-18; First posted 2011-01-19 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Sedentary Lifestyle; Obesity; General Well-being
Keywords: Behavioral economics; Incentives; Health
MeSH Terms: conditions — Sedentary Behavior; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Hold-out control (No Intervention): Hold-out control: participants will be asked to refrain from using the walkstations for the duration of the study (90 days).
- Personal incentive (Active Comparator): Personal incentive: Participants will receive $3 for each time they use the walkstation.
  Interventions: Behavioral: Incentives for walkstation usage
- Charitable incentive (Experimental): Charitable incentive: $3 will be donated to charity every time the participant uses the walkstation.
  Interventions: Behavioral: Incentives for walkstation usage

INTERVENTIONS:
Behavioral: Incentives for walkstation usage — The investigators are testing the effect of two different incentive schemes on people's usage of walkstations at work: either a personal incentive (in which people receive personal financial benefit for using the walkstations) vs. a charitable incentive (in which others receive financial benefit if a given individual uses the walkstation).
  Arms: Charitable incentive; Personal incentive

SUMMARY:
Employees of Blue Shield of California (BSC) will be recruited to participate to regularly use Walkstations. Some participants will be randomly assigned to a "hold out" control condition and the remainder will be assigned to one of two experimental treatments: Personal Incentive vs. Charitable Incentive. In the Personal Incentive condition people will be paid $3 for every completed Walkstation session, whereas for participants in the Charitable Incentive condition $3 will be donated to a specific charity. The incentives will operate for approximately 45 days and then for an additional 45 days participants in the two experimental conditions will have access to the Walkstations. Participants in the hold out control condition will begin using the Walkstations after the initial 90 day period.

ELIGIBILITY:
Inclusion Criteria:

* Must pass the ParQ

Exclusion Criteria:

* Ineligible if person did not pass ParQ AND did not provide doctor's note authorizing their participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-02; Primary Completion 2013-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Walkstation usage | 45 days

SECONDARY OUTCOMES:
Questionnaire | baseline; 45 days; 90 days
  Participants will be asked to complete a questionnaire that assesses job satisfaction, personal well-being, and health behaviors
Walkstation usage | 90 days
Biometrics | baseline & 45 days
  Height, weight, and blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Blue Shield of California, San Francisco, California, United States